CLINICAL TRIAL: NCT00733811
Title: Phase IV Study of the Use of Sequential DFP-DFO Versus DFP in Thalassemia Major Patients
Brief Title: Efficacy Study of the Use of Sequential DFP-DFO Versus DFP
Acronym: SEQDFPDFO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera V. Cervello (Other)
Responsible Party: Aurelio Maggio, AO V Cervello
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOVCervello
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-07

CONDITIONS: Beta-Thalassemia; Thalassemia Major
Keywords: thalassemia major; chelation treatment; secondary hemochromatosis
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferiprone; Isoflurophate; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sequential treatment including DFP at 75 mg/kg, divided into three oral daily doses, for four days per week and DFO by subcutaneous infusions (8-12h) at 50 mg/kg/day for the remaining three days per week
  Interventions: Drug: Deferiprone (DFP) and Deferoxamine (DFO)
- 2 (Active Comparator): Deferiprone alone at 75 mg/kg divided into three oral daily doses
  Interventions: Drug: Deferiprone (DFP)

INTERVENTIONS:
Drug: Deferiprone (DFP) and Deferoxamine (DFO) — Sequential treatment including DFP at 75 mg/kg for four days per week and DFO by subcutaneous infusions (8-12h) at 50mg/kg/day for the remaining three days per week
  Other Names: DFP (Apotex, Canada); DFO (Biofutura Pharma S.p.A.,Italy)
  Arms: 1
Drug: Deferiprone (DFP) — DFP alone at 75 mg/kg divided into three oral daily doses
  Other Names: DFP (Apotex, Canada)
  Arms: 2

SUMMARY:
Changes in chelation treatment and transfusion practices, during the past two decades, have dramatically improved the prognosis of thalassemia major patients.Deferiprone (DFP) has been compared with deferoxamine (DFO), using different schedules of treatment, in the majority of the 13 clinical trials published between 1990 and 2008.No statistically significant difference was shown between these two interventions during, at most, 18 months of treatment.Three randomised trials that compared sequential DFP-DFO treatment versus DFO alone reported controversial results but this could be due to small sample sizes and short treatment duration. In fact, no trial with treatment duration longer than 18 months15, which reported on mortality, adverse events, serum ferritin concentrations, as well as costs has so far been published.

This long-term sequential DFP-DFO treatment versus DFP alone treatment trial was conducted to assess the impacts of these chelation treatments on serum ferritin concentrations, mortality, adverse events, and costs in thalassemia major patients.

DETAILED DESCRIPTION:
The trial was designed as a multicentre randomised open-label trial with blinded data management and data analyses, to assess whether either treatment was superior to the other. The trial was performed on behalf of the Italian Society for the study of Thalassemia and Haemoglobinopathies (SoSTE). The investigators initiated, carried out, and controlled the trial, which was conducted without influence of the non-commercial sponsor.16

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia major patients with serum ferritin concentration between 800 to 3,000 ng/ml and were over 13 years of age

Exclusion Criteria:

* Known intolerance to one of the trial treatments
* Platelet count < 100,000/mm3 or or leukocyte count < 3,000/mm3
* Severe liver damage indicated by ascites
* Heart failure

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Actual)
Dates: Start 2000-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
difference between multiple observations of the serum ferritin concentrations | five-year treatment

SECONDARY OUTCOMES:
the difference between the T2* signal at magnetic resonance imaging (MRI) of heart and liver at T0 and T1 time (see below); survival analysis; adverse events; treatment failures; and costs. | five years

CONTACTS AND LOCATIONS:
Overall Officials: AURELIO MAGGIO, M.D., Study Chair — Azienda Ospedaliera V. Cervello
Locations (1):
- Ao V. Cervello, Palermo, Italy

REFERENCES:
- [Derived] Maggio A, Vitrano A, Capra M, Cuccia L, Gagliardotto F, Filosa A, Romeo MA, Magnano C, Caruso V, Argento C, Gerardi C, Campisi S, Violi P, Malizia R, Cianciulli P, Rizzo M, D'Ascola DG, Quota A, Prossomariti L, Fidone C, Rigano P, Pepe A, D'Amico G, Morabito A, Gluud C. Long-term sequential deferiprone-deferoxamine versus deferiprone alone for thalassaemia major patients: a randomized clinical trial. Br J Haematol. 2009 Apr;145(2):245-54. doi: 10.1111/j.1365-2141.2009.07609.x. Epub 2009 Feb 19. PMID 19236376